CLINICAL TRIAL: NCT06799910
Title: Optimization of Fluid Balance Guided by Bioelectrical Impedance Analysis in Patients Undergoing Continuous Renal Replacement Therapy in Critical Care
Acronym: OBHIMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0069
Record Dates: First submitted 2024-11-12; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Congestion; RRT; UF; Bio-impendance Analysis; Fluid Removal; Diuretics; Overload
Keywords: bio-impendance analysis; fluid removal; diuretics; overload; congestion; RRT; UF
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: A Pilot, Controlled, Open-Label, Randomized Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free UF Prescription (Active Comparator): Free UF Prescription :
  The UF (ml/h) is prescribed by the responsible physician based on the patient's clinical, congestive, and hemodynamic status. The physician can implement the UF whenever necessary based on the patient's hemodynamic condition.
  Interventions: Procedure: continuous renal replacement therapy (CRRT)
- UF Prescription Guided by the ECW/TBWat Ratio (Experimental): Experimental Group - UF Prescription Guided by the ECW/TBWat Ratio :
  * In the experimental group, the patient will receive a prescription for UF guided by the ECW/TBWat ratio. The goal is to achieve an ECW/TBWat ratio of less than 0.400 by the end of the 72-hour RRT session.
  * To meet this objective, the physician must measure the ECW/TBWat ratio each time the UF is adjusted. If the patient's ECW/TBWat ratio is less than 0.400 at the measurement time, the goal is to maintain it below 0.400 during the RRT session.
  * To calculate the ECW/TBWATratio, the Inbody BWA 2.0 device requires the initial TBW, which will be measured by the Hill-Room Acella 900 bed (Hill-Room, Batesville, USA).
  * The ratio is calculated by the Inbody BWA 2.0 and is based on the average of 3 consecutive measurements.
  * The physician determines the prescription for adjusting the UF (ml/h) based on the patient's hemodynamic and clinical condition during the RRT session.
  Interventions: Other: Free UF Prescription

INTERVENTIONS:
Procedure: continuous renal replacement therapy (CRRT) — The patient is included in the study once they meet the eligibility criteria and as soon as the responsible physician has prescribed RRT according to the department's protocol. Randomization will be performed, and the patient will be assigned to either the standard or experimental groups.
  Arms: Free UF Prescription
Other: Free UF Prescription — The UF (ml/h) is prescribed by the responsible physician based on the patient's clinical, congestive, and hemodynamic status. The physician can implement the UF whenever necessary based on the patient's hemodynamic condition.
  Arms: UF Prescription Guided by the ECW/TBWat Ratio

SUMMARY:
In critical care, hemodynamic instability often requires volume expansion to restore tissue perfusion, increasing fluid balance and TBW, factors associated with higher mortality. Excess fluid leads to organ dysfunction due to venous congestion, making fluid removal crucial. When diuretics fail, RRT, typically through continuous renal replacement therapy (CRRT), is recommended. However, prescribing the correct level of UF is challenging; insufficient UF can worsen edema, while excessive UF risks hemodynamic instability. This pilot, single-center, prospective, interventional, randomized, controlled, open-label study includes two parallel groups: a standard group with UF prescribed by the physician based on clinical and hemodynamic status and an experimental group with UF guided by the extracellular to total body water (ECW/TBWat) ratio measured by BIA. The aim is to determine if ECW/TBW-guided UF improves fluid and TBW reduction over a 72-hour RRT period.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* The patient was hospitalized in the intensive care unit of Amiens-Picardie University Hospital.
* Patient with an increase in fluid balance (TBW > 5%)
* Patient receiving continuous veno-venous hemofiltration (CVVH) on a PrismaFlexR or PrisMaxR machine, initiated due to oliguria, potassium level > 6.5 mmol/L, urea level > 25 mmol/L, or creatinine > 300 µmol/L and severe metabolic acidosis (pH < 7.2).
* Hemodynamically stable patient with a mean arterial pressure (MAP) > 65 mmHg for more than 4 hours with norepinephrine.
* Signed consent to participate in the study by the patient or, if unconscious, their legal representative/next of kin.

Exclusion Criteria:

* Invalid BIA measurements
* Internal device powered by an electrical current (pacemaker, implantable cardioverter-defibrillator, neurostimulator)
* Cardiac arrhythmia (atrial fibrillation, atrial flutter) present at the inclusion
* Chronic dialysis patient
* Moribund patient
* The patient is on extracorporeal mechanical support
* Hemorrhagic shock
* Pregnant woman
* Patient under guardianship or conservators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
comparison of TBW between both groups | at 72 hours
  To assess the impact of UF prescription guided by the ECW/TBWat ratio on weight loss, a comparison of TBW (∆TBW) between the two groups will be conducted. The ∆TBW is the difference between the initial TBW at H0 and the TBW at H72.

SECONDARY OUTCOMES:
Variation of cumulative net UF | at 72 hours
  The net UF is the difference between the fluids removed by RRT and the replacement fluids infused before and after the RRT filter. The cumulative net UF is the UF measured from H0 to H72. The volume of UF and infused replacement fluid will be calculated using data extracted from the memory card of the RRT machine.
Measurement of the net UF rate | at 72 hours
  Measurement of the net UF rate (ml/kg/h): The net UF rate is calculated as follows: cumulative net UF / (TBW at H0) x effective treatment duration during the 72 hours of the study. The treatment duration will be measured using data extracted from the memory card of the RRT machine.
Measurement of the ECW/TBWATratio and its association with the VeXUS score | day 0
  Measurement of the ECW/TBWATratio and its association with the VeXUS score at H0 . The VeXUS score is an echocardiographic score (ranging from 0 to 3) used to analyze venous congestion at the cardiac, renal, and hepatic levels.
Measurement of the ECW/TBWATratio and its association with the VeXUS score | at 72 hours
  Measurement of the ECW/TBWATratio and its association with the VeXUS score at H72 . The VeXUS score is an echocardiographic score (ranging from 0 to 3) used to analyze venous congestion at the cardiac, renal, and hepatic levels.
Measurement of the ECW/TBWAT ratio | day 0
  Measurement of the ECW/TBWATratio and its association with conventional right heart function parameters and those evaluated by speckle tracking at H0. The speckle tracking-based parameters used will measure: (a) Longitudinal displacement of the septal and lateral walls and right ventricular shortening; (b) Global longitudinal strain and free wall strain of the right ventricle and (c) Right atrial strain (reservoir, conduit, and contraction phases). The parameters will be measured offline using the QLAB 15.0 software (Philips Healthcare).
Measurement of the ECW/TBWAT ratio | 72 hours
  Measurement of the ECW/TBWATratio and its association with conventional right heart function parameters and those evaluated by speckle tracking at H72. The speckle tracking-based parameters used will measure: (a) Longitudinal displacement of the septal and lateral walls and right ventricular shortening; (b) Global longitudinal strain and free wall strain of the right ventricle and (c) Right atrial strain (reservoir, conduit, and contraction phases). The parameters will be measured offline using the QLAB 15.0 software (Philips Healthcare).
number of filters used in both groups | at 24 hours
  Reporting of complications related to RRT in both groups : number of filters used
number of filters used in both groups | at 48 hours
  Reporting of complications related to RRT in both groups : number of filters used
number of filters used in both groups | at 72 hours
  Reporting of complications related to RRT in both groups : number of filters used
duration of use for each filter in both groups | at 24 hours
  complications related to RRT in both groups : duration of use for each filter in both groups
duration of use for each filter in both groups | at 48 hours
  complications related to RRT in both groups : duration of use for each filter in both groups
duration of use for each filter in both groups | at 72 hours
  complications related to RRT in both groups : duration of use for each filter in both groups
Number of hypotensive episodes during dialysis | at 24 hours
  Number of hypotensive episodes during dialysis: A hypotensive episode is defined as a mean arterial pressure (MAP) < 65 mmHg for 1 minute, measured using hemodynamic monitoring
Number of hypotensive episodes during dialysis | at 48 hours
  Number of hypotensive episodes during dialysis: A hypotensive episode is defined as a mean arterial pressure (MAP) < 65 mmHg for 1 minute, measured using hemodynamic monitoring
Number of hypotensive episodes during dialysis | at 72 hours
  Number of hypotensive episodes during dialysis: A hypotensive episode is defined as a mean arterial pressure (MAP) < 65 mmHg for 1 minute, measured using hemodynamic monitoring
Number of arrhythmias in both groups | at 24 hours
  Number of arrhythmias in both groups
Number of arrhythmias in both groups | at 48 hours
  Number of arrhythmias in both groups
Number of arrhythmias in both groups | at 72 hours
  Number of arrhythmias in both groups
Number of arrhythmias with hemodynamic instability | at 24 hours
  Number of arrhythmias with hemodynamic instability
Number of arrhythmias with hemodynamic instability | at 48 hours
  Number of arrhythmias with hemodynamic instability
Number of arrhythmias with hemodynamic instability | at 72 hours
  Number of arrhythmias with hemodynamic instability
Measurement of serum potassium | at 24 hours
  Measurement of serum potassium
Measurement of serum potassium | at 48 hours
  Measurement of serum potassium
Measurement of serum potassium | at 72 hours
  Measurement of serum potassium
Measurement of serum phosphate | at 24 hours
  Measurement of serum phosphate
Measurement of serum phosphate | at 48 hours
  Measurement of serum phosphate
Measurement of serum phosphate | at 72 hours
  Measurement of serum phosphate
Cumulative volume of crystalloid administration | at 72 hours
  Cumulative volume of crystalloid administration
Cumulative volume of colloid administration | at 72 hours
  Cumulative volume of colloid administration
Cumulative dose of norepinephrine administration | at 72 hours
  Cumulative dose of norepinephrine administration
Duration of norepinephrine administration | at 72 hours
  Duration of norepinephrine administration
Duration of mechanical ventilation | at day 30
  Duration of mechanical ventilation
30-day mortality | at day 30
  30-day mortality
Length of stay in intensive care | at day 30
  Length of stay in intensive care
Length of stay at the hospital | at day 30
  Length of stay at the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No